CLINICAL TRIAL: NCT04419025
Title: Determination of Efficacy of N-Acetylcysteine in Preventing Those With Mild or Moderate COVID-19 From Progressing to Severe Disease
Brief Title: Efficacy of N-Acetylcysteine (NAC) in Preventing COVID-19 From Progressing to Severe Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Responsible Party: Principal Investigator, Melisa Lai-Becker, Chief, CHA Everett Hospital Emergency Department; Director, CHA Division of Medical Toxicology, Cambridge Health Alliance
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHA-IRB-1139/05/20
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: COVID; Sars-CoV2; SARS-Associated Coronavirus as Cause of Disease Classified Elsewhere; Oxidative Stress
Keywords: Glutathione; Acetylcysteine; Oxidative stress; NAC; COVID; COVID-19; SARS-CoV2
MeSH Terms: conditions — COVID-19 | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study.
  One arm is the intervention arm - those receiving N-acetylcysteine (NAC). One arm is the control group - those not receiving N-acetylcysteine (NAC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NAC (Active Comparator): Patients receiving N-acetylcysteine (NAC)
  Interventions: Drug: N-acetylcysteine
- Control (No Intervention): Patients not receiving N-acetylcysteine (NAC)

INTERVENTIONS:
Drug: N-acetylcysteine — Oral formulation: 600 mg capsules of N-acetylcysteine
  Other Names: NAC, acetylcysteine, N-acetyl-L-cysteine, NALC
  Arms: NAC

SUMMARY:
The purpose of this study is to assess the efficacy of N-acetylcysteine (NAC) in preventing those with mild or moderate COVID-19 from progressing to severe disease

DETAILED DESCRIPTION:
After being informed of the study and potential risks and benefits, patients meeting eligibility requirements will be randomized to receive oral N-acetylcysteine (NAC) as follows:

Inpatients:

* N-acetylcystine (NAC) 25 mg/kg PO (rounded up to the nearest 600 mg) q4hrs until discharge
* N-acetylcysteine (NAC) 1200 mg PO BID x 1 week post-discharge

Outpatients:

- N-acetylcysteine (NAC) 2400 mg PO x 1 then 1200 mg PO BID x 2 weeks

ELIGIBILITY:
Inclusion Criteria:

* known or suspect COVID-19 disease AND one or more of the following influenza-like symptoms, including: diarrhea vomiting fever (subjective or measured) chills myalgias fatigue sore throat headache cough nasal/sinus congestion or rhinorrhea shortness of breath chest pain

Exclusion Criteria:

* Minors, pregnant women and people unable to provide informed consent are excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Decrease in Respiratory Rate | First hour after first dose of NAC
  Decrease in dyspnea measured by respiratory rate (RR)
Hospital length of stay (LOS) | Through study completion, average 9 months
  Hospital LOS for admitted patients
Need for mechanical ventilation | Through study completion, average 9 months
  Whether a patient needed mechanical ventilation (intubation)
Length of time intubated | Through study completion, average 9 months
  If intubated, how long needing mechanical ventilation
Need for hospitalization | Through study completion, average 9 months
  Outpatients on NAC needing admission to the hospital
Recovery disposition | Through study completion, average 9 months
  Whether outpatients continued to recover as outpatients; whether admitted patients were managed on medical floors or level of care increased to ICU level of care; whether patients expired

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - CHA Cambridge Hospital, Cambridge, Massachusetts
  - CHA Everett Hospital, Everett, Massachusetts
  - CHA Respiratory Clinic, Somerville, Massachusetts
  - CHA Somerville campus, Somerville, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Information that underlies results in published data
Supporting Information: Study Protocol, ICF
Time Frame: Six months after publication available for a year
Access Criteria: Written request; to be reviewed by the PI
URL: http://www.NACinCOVID.info

REFERENCES:
- See also: Website reviewing reasoning and references for using NAC as adjuvant therapy in treatment of COVID-19 — http://www.NACinCOVID.info
- See also: Website reviewing reasoning and references for using NAC as adjuvant therapy in treatment of COVID-19 — http://www.NACinCOVID.net
- See also: Website reviewing reasoning and references for using NAC as adjuvant therapy in treatment of COVID-19 — http://www.NACinCOVID.org